CLINICAL TRIAL: NCT04092114
Title: Community Health Clinic Model for Agency in Relationships and Safer Microbicide Adherence (CHARISMA) Expansion Study
Brief Title: CHARISMA Expansion Study
Acronym: CHARISMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: Wits Reproductive Health and HIV Institute (Other); FHI 360 (Other); United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AID-OAA-A-15-00032
Record Dates: First submitted 2019-05-28; First posted 2019-09-17 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Relationship Dynamics; Pre-exposure Prophylaxis (PrEP) Adherence
Keywords: PrEP (Pre-exposure Prophylaxis); HIV prevention; Intimate Partner Violence (IPV)

STUDY DESIGN:
Intervention Model Description: Two-arm, randomized (1:1), controlled study of a behavioral intervention to increase adherence to daily oral PrEP, improve partner relationships (communication and support) and reduce social harms and IPV.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): Receives Standard of Care (SOC) services established in accordance with the South African Department of Health (DoH) PrEP (Pre-exposure Prophylaxis) guidelines.
  Interventions: Other: Control
- CHARISMA Intervention (Experimental): Receives SOC (Standard of care) per control arm plus provider-administration of HEART (HEAlthy Relationship Assessment Tool) and provider-administration of CHARISMA (the Community Health clinic model for Agency in Relationships and Safer Microbicide Adherence) counseling modules, as applicable:
  * Module A: General Partner Communication and Relationship Skills
  * Module B: Partner Disclosure and Communication around PrEP Use
  * Module C: Responding to Intimate Partner Violence and Safety Planning
  Interventions: Behavioral: CHARISMA Intervention

INTERVENTIONS:
Other: Control — Standard of care (SOC) HIV prevention services in line with the South African DoH (Department of Health) PrEP (Pre-exposure Prophylaxis) rollout program that include daily oral TDF/FTC (tenofovir disoproxil fumarate/emtricitabine). In addition, risk reduction counseling, IPV (Intimate Partner Violence) screening using the VAWS (WHO Violence Against Women Survey) with referrals for counseling, medical care, or shelter assistance, among other care options, if needed and an informational packet regarding HIV prevention services for themselves and male partners will be offered
  Arms: Control
Behavioral: CHARISMA Intervention — SOC (Standard of Care) per control arm plus provider-administration of HEART and provider-administration of CHARISMA counseling modules, as applicable:
  * Module A: General Partner Communication and Relationship Skills
  * Module B: Partner Disclosure and Communication around PrEP Use
  * Module C: Responding to Intimate Partner Violence and Safety Planning
  Arms: CHARISMA Intervention

SUMMARY:
The CHARISMA Expansion Study is a two-arm, randomized (1:1), controlled study of a behavioral intervention-the Community Health clinic model for Agency in Relationships and Safer Microbicide Adherence (CHARISMA)-to reduce social harms (SHs) and intimate partner violence (IPV), increase healthy relationship dynamics and oral PrEP (pre-exposure prophylaxis) TDF/FTC (tenofovir disoproxil fumarate/emtricitabine), hereafter called PrEP, adherence among enrolled women. This study is an expansion of the CHARISMA intervention pilot study which was appended to the Microbicide Trials Network (MTN)-025 HOPE (HIV Open Label Prevention Extension) study.

CHARISMA is defined by the use of a tool, called the CHARISMA HEAlthy Relationship Assessment Tool (HEART) used in combination with three counselling modules:

* Module A: General Partner Communication and Relationship Skills
* Module B: Partner Disclosure and Communication around PrEP Use
* Module C: Responding to Intimate Partner Violence and Safety Planning

DETAILED DESCRIPTION:
The CHARISMA Expansion Study is a two-arm, randomized (1:1), controlled study of a behavioral intervention-the Community Health clinic model for Agency in Relationships and Safer Microbicide Adherence (CHARISMA)-which aims to reduce social harms (SHs) and intimate partner violence (IPV), increase healthy relationship dynamics and oral PrEP TDF/FTC (hereafter called PrEP) adherence among enrolled women. This study is an expansion of the CHARISMA intervention pilot study which was appended to the Microbicide Trials Network (MTN)-025 HOPE study and will conclude in 2018.

CHARISMA is defined by the use of a tool, called the CHARISMA HEAlthy Relationship Assessment Tool (HEART) used in combination with three counselling modules:

* Module A: General Partner Communication and Relationship Skills
* Module B: Partner Disclosure and Communication around PrEP Use
* Module C: Responding to Intimate Partner Violence and Safety Planning

The HEART will be used to assess the status of women's relationships and experience of IPV in the intervention arm. The HEART, previously piloted in HOPE, is a tool used to facilitate assessment of, and response to, the range of positive and negative effects of HIV prevention product use experienced by women in intimate partner relationships.

In September 2015, the World Health Organization issued guidelines recommending PrEP be offered to all persons at substantial HIV risk (defined as HIV incidence rate above 3%) worldwide. In sub-Saharan Africa, women account for 58% of the total number of people living with HIV. Given the high HIV incidence and evidence for high potential effectiveness of PrEP when adherence to product use is high, PrEP delivery, adherence, and associated male partner dynamics should be evaluated among a broad age range of women.

This study will enroll sexually active, HIV-uninfected women, who are trial naïve, non-pregnant and aged 18-45 years (inclusive). PrEP, delivered according to national guidelines, IPV screening using the WHO Violence Against Women Survey (VAWS) and referrals for care will be offered to all eligible participants as Standard of Care (SOC) in the control arm. CHARISMA intervention arm participants will receive in-person counselling as part of the CHARISMA intervention to help them assess and build support for PrEP use within their relationships. SHs, IPV, relationship dynamics (e.g. communication, support) and PrEP adherence will be compared across the two arms. Social harms are defined as non-clinical trial related adverse events that result in psychosocial, social, or physical harm among women.

Design: Two-arm, randomized (1:1), controlled study of a behavioral intervention to increase adherence to daily oral PrEP, improve partner relationships (communication and support) and reduce SH and IPV.

A PrEP delivery project will be established in accordance with national guidelines in South African Department of Health (DoH) PrEP guidelines supplemented by the addition of the CHARISMA intervention. Participants presenting for enrolment will be randomized to one of two study arms below:

1. Control: Standard of care (SOC) HIV prevention services in line with the South African DoH PrEP rollout program that include daily oral TDF/FTC. In addition, risk reduction counseling, IPV screening using the VAWS with referrals for counseling, medical care, or shelter assistance, among other care options if needed and an informational packet regarding HIV prevention services for themselves and male partners will be offered;
2. CHARISMA Intervention: SOC per control arm plus provider-administration of HEART and provider-administration of CHARISMA counseling modules, as applicable:

   * Module A: General Partner Communication and Relationship Skills
   * Module B: Partner Disclosure and Communication around PrEP Use
   * Module C: Responding to Intimate Partner Violence and Safety Planning

Population: Approximately four hundred sexually active, HIV-uninfected women who are trial naïve, non-pregnant, and not planning to be pregnant for the next six months, non-breastfeeding, aged 18 to 45 years of age (inclusive)

Study Site(s): Wits RHI (Reproductive Health and HIV Institute) Clinical Research Site, Johannesburg, South Africa Other site(s) to be determined

Approach: This project will offer a PrEP delivery package within two arms of a controlled, randomized study of women to evaluate the impact of the CHARISMA intervention when paired with PrEP delivery.

Study Duration: Accrual will require approximately 12 months. Each participant presenting for PrEP education and services will be enrolled and followed for 6 months. Participants in both study arms will participate in scheduled visits for screening, enrollment, and months 1, 3, and 6 of follow-up. A subset of participants will be asked to participate in a qualitative interview at month 6, and/or month 9.

Primary Objectives:

1. To determine the effectiveness of the CHARISMA intervention in increasing PrEP adherence/persistence at month 6;
2. To determine the effectiveness of the CHARISMA intervention in reducing reported experiences of social harms while on PrEP;
3. To determine the effectiveness of the CHARISMA intervention in reducing reported experiences of IPV (irrespective of time on PrEP);
4. To determine the effectiveness of CHARISMA on participant's reported relationship dynamics, including disclosure of PrEP use, support for product use, and communication;

   Secondary Objective:
5. To explore the acceptability and feasibility of the CHARISMA intervention; and

Exploratory Objective:

7) To assess the sensitivity and specificity of a brief IPV screening tool compared to a longer validated tool in identifying cases of IPV.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide written informed consent and locator information
* Reports having a current male primary partner,
* Sexually active, defined by vaginal intercourse with a male at least 4 times per month in the past 3 months and plan to be sexually active during the study duration
* Not pregnant (defined by urine pregnancy testing) and not breastfeeding
* Not planning on becoming pregnant in the next 6 months
* English or Zulu speaking
* HIV negative based on negative HIV rapid tests, at the time of enrollment

Exclusion Criteria:

* Previously participated in a clinical trial or a longitudinal HIV prevention research study
* Unwilling to use daily oral PrEP
* Has any significant medical condition or other condition that, in the opinion of the Principal Investigator (PI)/designee, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 407 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2020-05-25 (Actual); Study Completion 2020-05-25 (Actual)

PRIMARY OUTCOMES:
PrEP adherence/persistence by measurement | 3 months
  Adherence will be ascertained through measurement of TFV-DP (tenofovir-diphosphate) in dried blood spot (DBS) specimens. DBS collected via blood draw at Month 3 and 6 follow-up visits will be used for retrospective PCR testing for tenofovir levels (although DBS is collected at Enrollment and Month 1 as well).
PrEP adherence/persistence by measurement | 6 months
  Adherence will be ascertained through measurement of TFV-DP in DBS specimens. DBS collected via blood draw at Month 3 and 6 follow-up visits will be used for retrospective PCR testing for tenofovir levels (although DBS is collected at Enrollment and Month 1 as well).
PrEP adherence/persistence by self-report | 3 months
  Self-reported data on PrEP adherence will be collected via standardized questionnaires to better understand patterns of PrEP use and reasons for poor adherence or discontinuation. The tool used for the assessment is the WHO Violence Against Women Survey (VAWS). VAWS consists of behavior-specific items related to psychological (four items), physical (six items) and sexual violence (three items). The physical violence items are further divided into 'moderate' (the two first items) and 'severe' (the following four items) violence based on the likelihood of physical injury. Values are considered worse as responses to experiences of violence increase from no=0, to one=1, few=2, and many=3 times.
PrEP adherence/persistence by self-report | 6 months
  Self-reported data on PrEP adherence will be collected via standardized questionnaires to better understand patterns of PrEP use and reasons for poor adherence or discontinuation. The tool used for the assessment is the WHO VAWS. VAWS consists of behavior-specific items related to psychological (four items), physical (six items) and sexual violence (three items). The physical violence items are further divided into 'moderate' (the two first items) and 'severe' (the following four items) violence based on the likelihood of physical injury. Values are considered worse as responses to experiences of violence increase from no=0, to one=1, few=2, and many=3 times.
Incidence of social harms (SHs) using a SHs questionnaire | Anytime during the study, up to 6 months
  SH in this study could include negative consequences related to study participation, PrEP use disclosure, stigma, gender-based violence, and relationship problems. Participants will be screened for SH resulting from product use or study participation at Enrollment, Month 3, and Month 6, and may report a social harm to staff at any time during the study.
IPV: Self-report of a) any IPV or b) physical or sexual IPV during study participation. | Anytime during the study, up to 6 months
  All participants will receive SOC IPV screening at enrollment and at the Month 3 and Month 6 visits and may report IPV to staff at any time during the study. SOC IPV screening will include clinical screening with a validated IPV measurement tool-the WHO VAWS. The WHO considers the VAWS to be a valid and reliable measure of GBV (gender-based violence) and is therefore a reasonable SOC screening tool for this study.
Percent of participants who disclosed PrEP product use to a partner, which is reported via a questionnaire | Enrollment
  Consistent with the primary objective to determine the effect of CHARISMA on participants' relationship dynamics, the following endpoints will be assessed:
  * Disclosure of PrEP use to male partners: Self-report that participants have told their partners that they are using PrEP
  * Male partner support for product use: Self-report that male partners support or accept (i.e. do not oppose) their PrEP use
  * Communication with male partners: Self-report of partnership communication dynamics.
  All participants will be asked about relationship dynamics, including disclosure of PrEP use, support for product use, and communication during enrollment, month 3, and 6 follow-up visits, and as needed during month 1 visits.
Percent of participants who disclosed PrEP product use to a partner, which is reported via a questionnaire | 1 month
  Consistent with the primary objective to determine the effect of CHARISMA on participants' relationship dynamics, the following endpoints will be assessed:
  * Disclosure of PrEP use to male partners: Self-report that participants have told their partners that they are using PrEP
  * Male partner support for product use: Self-report that male partners support or accept (i.e. do not oppose) their PrEP use
  * Communication with male partners: Self-report of partnership communication dynamics All participants will be asked about relationship dynamics, including disclosure of PrEP use, support for product use, and communication during enrollment, month 3, and 6 follow-up visits, and as needed during month 1 visits.
Percent of participants who disclosed PrEP product use to a partner, which is reported via a questionnaire | 3 months
  Consistent with the primary objective to determine the effect of CHARISMA on participants' relationship dynamics, the following endpoints will be assessed:
  * Disclosure of PrEP use to male partners: Self-report that participants have told their partners that they are using PrEP
  * Male partner support for product use: Self-report that male partners support or accept (i.e. do not oppose) their PrEP use
  * Communication with male partners: Self-report of partnership communication dynamics All participants will be asked about relationship dynamics, including disclosure of PrEP use, support for product use, and communication during enrollment, month 3, and 6 follow-up visits, and as needed during month 1 visits.
Percent of participants who disclosed PrEP product use to a partner, which is reported via a questionnaire | 6 months
  Consistent with the primary objective to determine the effect of CHARISMA on participants' relationship dynamics, the following endpoints will be assessed:
  * Disclosure of PrEP use to male partners: Self-report that participants have told their partners that they are using PrEP
  * Male partner support for product use: Self-report that male partners support or accept (i.e. do not oppose) their PrEP use
  * Communication with male partners: Self-report of partnership communication dynamics All participants will be asked about relationship dynamics, including disclosure of PrEP use, support for product use, and communication during enrollment, month 3, and 6 follow-up visits, and as needed during month 1 visits.

SECONDARY OUTCOMES:
Acceptability and feasibility assessed by intervention tool utilization as reported in response to a questionnaire".- | 6 months
  Consistent with the secondary objective to explore the acceptability and feasibility of CHARISMA, the following endpoint will be assessed:
  • Acceptability: Participant ranking of intervention components
Acceptability and feasibility assessed by participants' accounts of utilizing the CHARISMA intervention, as reported during an interview. | 6 months
  Consistent with the secondary objective to explore the acceptability and feasibility of CHARISMA, the following endpoint will be assessed:
  • Acceptability: Participant qualitative report via interview
Acceptability and feasibility assessed by participants' accounts of utilizing the CHARISMA intervention, as reported during an interview. | 9 months
  Consistent with the secondary objective to explore the acceptability and feasibility of CHARISMA, the following endpoint will be assessed:
  • Acceptability: Participant qualitative report via interview
Feasibility of the CHARISMA intervention - Time to completion | Anytime during the study, up to 6 months
  Consistent with the secondary objective to explore the acceptability and feasibility of CHARISMA, the following endpoint will be assessed:
  • Feasibility: Process indicator of time to completion.
Percentage of participants who complete the intervention as outlined by the protocol, assessed via case report forms | Anytime during the study, up to 6 months
  Consistent with the secondary objective to explore the acceptability and feasibility of CHARISMA, the following endpoint will be assessed:
  • Feasibility: Process indicator of intervention fidelity
Feasibility of the CHARISMA intervention - Measure of surveys and modules completed | Anytime during the study, up to 6 months
  Consistent with the secondary objective to explore the acceptability and feasibility of CHARISMA, the following endpoint will be assessed:
  • Feasibility: Process indicator of percentage of surveys and modules completed
Feasibility of the CHARISMA intervention - Percentage of missing data | Anytime during the study, up to 6 months
  Consistent with the secondary objective to explore the acceptability and feasibility of CHARISMA, the following endpoint will be assessed:
  • Feasibility: Process indicator of percentage of missing HEART data.
Sensitivity and specificity of a brief intimate partner violence (IPV) screening tool compared to a longer validated tool in identifying cases of IPV. | 3 months
  All participants will receive IPV screening at enrollment and at the Month 3 and Month 6 visits. SOC IPV screening will include clinical screening with a validated IPV measurement tool-the WHO VAWS. The WHO considers the VAWS to be a valid and reliable measure of GBV and is therefore a reasonable SOC screening tool for this study.
Sensitivity and specificity of a brief IPV screening tool compared to a longer validated tool in identifying cases of IPV. | 6 months
  All participants will receive IPV screening at enrollment and at the Month 3 and Month 6 visits. SOC IPV screening will include clinical screening with a validated IPV measurement tool-the WHO VAWS. The WHO considers the VAWS to be a valid and reliable measure of GBV and is therefore a reasonable SOC screening tool for this study.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Montgomery, PhD, MHS, Principal Investigator — RTI International; Thesla Palanee, MMedSci,PhD,MSc, Principal Investigator — Wits RHI
Locations (1):
- Wits Reproductive Health and HIV Institute (Wits RHI), Johannesburg, South Africa

IPD SHARING:
Plan to Share IPD: No